CLINICAL TRIAL: NCT05255822
Title: Phase 2a Study in Healthy Adult Participants Pre-treated With INNA-051 and Challenged With Influenza Virus
Brief Title: INNA-051 Influenza Challenge Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ENA Respiratory Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INNA-051-IAV-HC-01
Record Dates: First submitted 2022-01-27; First posted 2022-02-25 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Influenza Prophylaxis
MeSH Terms: interventions — INNA-051

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INNA-051 arm 1 (Experimental): INNA-051 intranasal spray low dose administered once on each of Days -4 and -2 prior to viral challenge
  Interventions: Drug: INNA-051
- INNA-051 arm 2 (Experimental): NNA-051 intranasal spray high dose administered once on each of Days -4 and -2 prior to viral challenge
  Interventions: Drug: INNA-051
- Placebo (Placebo Comparator): Placebo intranasal spray low dose administered once on each of Days -4 and -2 prior to viral challenge
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: INNA-051 — Liquid for intra-nasal administration
  Arms: INNA-051 arm 1; INNA-051 arm 2
Other: Placebo — Liquid for intra-nasal administration
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled study of INNA-051 in healthy adults, administered prior to administration of an influenza challenge virus. This study will evaluate 2 active dose levels of INNA-051 and placebo.

DETAILED DESCRIPTION:
Healthy participants will be administered 2 doses on INNA-051 intra-nasally and subsequently administered influenza virus as a challenge. Participants will be quarantined for 8 days. Study assessments will be performed during this period and they will monitored for symptoms of influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* 18 to 55 years (inclusive) at time of consent
* In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety
* Agree to use highly effective contraception

Exclusion Criteria:

* History of, or currently active, symptoms or signs suggestive of URT or lower respiratory tract (LRT) infection within 4 weeks prior to the first study visit
* Any history or evidence of any other clinically significant or currently active systemic comorbidities including psychiatric disorders (includes participants with a history of depression and/or anxiety)
* Participants who have smoked ≥10 pack years at any time
* A total body weight ≤50 kg or body mass index (BMI) ≤18 kg/m2 or ≥35kg/m2.
* Pregnant or breast feeding
* Any significant abnormality altering the anatomy of the nose or nasopharynx that may interfere with the nasal assessments or viral challenge, clinically significant history of epistaxis, or any nasal or sinus surgery within 3 months of the first study visit
* vaccinations within the 4 weeks prior to the planned date of first dosing with IMP (10 days for SARS-CoV-2 vaccines, 6 months for influenza vaccine), or during the study
* Receipt of blood or blood products, or loss (including blood donations) of 470 mL or more of blood during the 3 months prior to dosing or planned in 3 months post.
* Receipt of any investigational product within 3 months (or 5 half-lives of the investigational product used in the other study, whichever is greater) prior to first dose with IMP, or 3 IMPs within prior 12 months, or prior administration with a virus from the same virus family as the challenge virus, or prior participation in another respiratory viral challenge study in the preceding 3 months
* Confirmed positive test for drugs of abuse or cotinine, history or presence of alcohol addiction, or excessive consumption of xanthine-containing substances
* A forced expiratory volume in 1 second (FEV1) <80%
* Positive HIV-1 or HIV-2 test, or positive test for hepatitis B or C

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Evaluate the antiviral effect of INNA-051 compared to placebo against influenza virus | To Day 8
  Change in total viral load area under the curve (AUC) measured by quantitative reverse transcriptase-polymerase chain reaction (qRT PCR) in treated participants vs. placebo participants.

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events | To Day 8
  Treatment emergent adverse events in INNA-051 arms compared to placebo
To evaluate the antiviral effect of INNA-051 in reducing viral load when compared to placebo | To Day 8
  * measurement of influenza viral load and duration of quantifiable measurements in nasopharyngeal swabs by qRT-PCR
  * Duration of quantifiable qRT-PCR measurements
To evaluate the antiviral effect of INNA-051 in reducing detectable virus levels when compared to placebo | To Day 8
  - Duration of quantifiable qRT-PCR measurements
To evaluate the antiviral effect of INNA-051 in reducing incidence of infection when compared to placebo | To Day 8
  Incidence of 2 quantifiable qRT PCR samples on 2 consecutive days
To evaluate the antiviral effect of INNA-051 in reducing symptoms of influenza infection when compared to placebo | To Day 8
  All symptoms will be self-reported by participants on a symptom diary card

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Parker, MD, Principal Investigator — Hvivo
Locations (1):
- hVIVO, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No